CLINICAL TRIAL: NCT07249476
Title: ENKLA-M : Study of NK Cells in the Monitoring of Patients With Acute Leukemia or Myelodysplasia
Brief Title: Study of NK Cells in the Monitoring of Patients With Acute Leukemia or Myelodysplasia
Acronym: ENKLA-M
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: EFS CPDL: French Blood Establishment Centre-Pays de la Loire (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC25_0333; ANSM - IDRCB (Other: 2025-A01929-40)
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Leukaemia (Acute Myeloid); Leukaemia (Acute Lymphoblastic); Myelodysplastic Syndrome
Keywords: VIDAZA; CSH graft; haematopoietic stem cell; natural killer cells; NK Cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Myelodysplastic Syndromes | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Additional blood and bone marrow samples will only be taken if a blood and/or bone marrow sample is planned during treatment and no additional blood or bone marrow punctures are performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AZA/DLI Group: > 20 Acute myeloid leukaemia/myelodysplastic syndrome patients receiving a matched transplant: 10 patients receiving AZA/DLI for relapse prevention. 10 patients not receiving AZA/DLI (control group).
  This group is monitored at diagnosis and for 12 months after transplantation.
  Interventions: Other: Bone marrow sampling (during routine care); Other: Blood samples (during routine care)
- Group without AZA/DLI: > 20 Acute myeloid leukaemia/myelodysplastic syndrome patients receiving a haploidentical transplant: 10 patients receiving AZA/DLI for relapse prevention. 10 patients not receiving AZA/DLI (control group).
  This group is monitored at diagnosis and for 12 months after transplantation.
  Interventions: Other: Bone marrow sampling (during routine care); Other: Blood samples (during routine care)
- LAL (Acute lymphoblastic leukaemia): 10 Patients with a (Acute lymphoblastic leukaemia).
  This group is monitored at diagnosis only.
  Interventions: Other: Bone marrow sampling (during routine care); Other: Blood samples (during routine care)

INTERVENTIONS:
Other: Bone marrow sampling (during routine care) — Bone marrow sample (1 ml)
Other: Blood samples (during routine care) — 3 tubes of 10 ml per visit

SUMMARY:
The aim of the ENKLA-M study is to collect samples from patients with acute Myeloid Leukemia (AML), Acute Lymphocytic Leukemia (ALL), and myelodysplastic syndrome (MDS) to study the evolution of blast phenotype (NK receptor ligands and adhesion molecules) and the biology of patients' NK cells). To do this, blood and bone marrow samples will be collected from patients at diagnosis in order to characterize: (I) the phenotype of ALL and AML blasts with respect to NK receptor ligands and adhesion molecules; (II) the phenotypic profile of NK cells, (III) to further characterize the NK cell repertoire dynamics over time (day 30, day 60, day 90, 6 months, and 1 year), focusing on NK cell populations identified in healthy individuals as particularly effective against leukemia, by defining their phenotypic and transcriptomic profiles; and (IV) the impact of azacitidine (AZA) and donor lymphocyte infusions (DLI) on the biology of NK cells in transplanted patients. Clinical data and KIR/HLA genetic profiles will be used to analyze all NK phenotypic and functional data, with the aim of better defining: (i) the key molecular interactions between NK cells and leukemic cells; (ii) markers of NK cell anti-leukemic efficacy during hematopoietic reconstitution; and (iii) whether AZA/DLI treatment enhances the functional potential of NK cells via KIR-HLA interaction, thereby improving their effectiveness against residual disease.

ELIGIBILITY:
INCLUSION CRITERIA

* Adult patients diagnosed with acute myeloid leukaemia (LAM), acute lymphoblastic leukaemia (LAL) or myelodysplastic syndrome (SMD).
* Adult patients receiving a HSC transplant.
* Adult patients receiving or not AZA treatment after transplantation.
* Patients who have signed a consent form.
* Patients affiliated with a social security system. EXCLUSION CRITERIA
* Minors,
* Pregnant and/or breastfeeding women
* Adult patients under guardianship,
* Protected persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with AML, ALL or MDS treated in the haematology department of Nantes University Hospital.
  The number of transplants performed for these conditions in the department suggests that 55 patients could be recruited at diagnosis (30 LAM patients, 10 LAL patients and 15 SMD patients).
  Among the LAM and SMD patients (n=45), we will identify 40 patients for post-transplant studies:
  >20 LAM/SMD patients receiving a matched transplant:
  * 10 patients receiving AZA/Donor Lymphocyte Injection for relapse prevention.
  * 10 patients not receiving AZA/Donor Lymphocyte Injection (control group). >20 LAM/SMD patients receiving a haploidentical transplant:
  * 10 patients receiving AZA/Donor Lymphocyte Injection for relapse prevention.
  * 10 patients not receiving AZA/Donor Lymphocyte Injection (control group).
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Define the KIR and HLA genetic markers associated with an anti-leukaemic response mediated by NK cells at different stages in the progression of Acute lymphocytic leukaemia or a myalodysplasia syndrome. | 12 months

SECONDARY OUTCOMES:
Assess the functional potential of different NK cell populations at diagnosis of acute myeloid leukaemia, acute lymphoblastic leukaemia and myelodysplastic syndrome (at each possible relapse of the patient). | 12 months
Assess NK cell reconstitution during transplant of hematopoietic stem cells. | 12 months
Assess the impact of the hypomethylating agent AZA used to prevent relapse after allogeneic transplantation for acute myeloid leukaemia or myelodysplastic syndrome on NK cells. | 12 months
Assess the impact of Donor Lymphocyte Injection used in the prevention of post-allogeneic transplant relapse on NK cells. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrice CHEVALLIER, Principal Investigator — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: Undecided